CLINICAL TRIAL: NCT02963935
Title: Effect and Safety of Liraglutide 3.0 mg as an Adjunct to Intensive Behaviour Therapy for Obesity in a Non-specialist Setting
Acronym: SCALE™ IBT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4274; U1111-1177-5059 (Other: World Health Organization (WHO))
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide; Behavioral: CMS Intensive Behavior Therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo; Behavioral: CMS Intensive Behavior Therapy

INTERVENTIONS:
Drug: liraglutide — Administered subcutaneously (s.c., under the skin) once daily for 56 weeks. Dose gradually increased to 3.0 mg
  Arms: Liraglutide
Drug: placebo — Administered subcutaneously (s.c., under the skin) once daily for 56 weeks. Dose gradually increased to 3.0 mg
  Arms: Placebo
Behavioral: CMS Intensive Behavior Therapy — Intensive Behaviour Therapy for obesity

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of the trial is to investigate the effect and safety of liraglutide 3.0 mg as an adjunct to intensive behaviour therapy for obesity in a non-specialist setting (IBT-CMS: Intensive Behaviour Therapy for obesity in a primary care setting according to Centers for Medicare & Medicaid Services (CMS) visit schedule).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* BMI above or equal to 30 kg/m^2
* Male or female, age 18 years or older at the time of signing informed consent

Exclusion Criteria:

* HbA1c (glycosylated haemoglobin) above or equal to 6.5% (at screening visit), or diagnosis of type 1 or type 2 diabetes mellitus
* Recent history of cardiovascular disease (myocardial infarction or stroke within the past 6 months), severe congestive heart failure (NYHA class III, IV), or second degree or greater heart block
* Personal or family history of Medullary Thyroid Carcinoma (MTC), or Multiple Endocrine Neoplasia type 2 (MEN2)
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice)
* Use in past 90 days of medications known to induce significant weight loss (e.g., prescription weight loss medications) or weight gain (e.g., chronic use of oral steroids, second generation antipsychotics)
* History of pancreatitis (acute or chronic)
* History of major depressive disorder within the past 2 years
* Any lifetime history of a suicide attempt
* Inadequately treated blood pressure defined as Grade 3 hypertension or higher (Systolic above or equal to 180 mmHg or diastolic above or equal to 110 mmHg)
* History of malignancy (except for non-melanoma skin cancer) within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/

REFERENCES:
- [Result] Wadden TA, Tronieri JS, Sugimoto D, Lund MT, Auerbach P, Jensen C, Rubino D. Liraglutide 3.0 mg and Intensive Behavioral Therapy (IBT) for Obesity in Primary Care: The SCALE IBT Randomized Controlled Trial. Obesity (Silver Spring). 2020 Mar;28(3):529-536. doi: 10.1002/oby.22726. PMID 32090517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 17 sites in the United States.
Pre-assignment Details: All the subjects received Intensive Behaviour Therapy (IBT) for obesity in a primary care setting according to Centers for Medicare & Medicaid Services (CMS) visit schedule during the trial.
Groups:
- Liraglutide 3.0 mg: Subjects received liraglutide 3.0 mg once daily by subcutaneous injection (in the abdomen, thigh or upper arm) irrespective of the timing of meals. Subjects received 0.6 mg liraglutide during the first week. The dose was escalated in weekly increments of 0.6 mg until they reached a maintenance dose of 3.0 mg after 4 weeks. The treatment period was 56 weeks. Subjects were also on CMS-IBT during the trial.
- Placebo: Subjects received matching placebo once daily by subcutaneous injection (in the abdomen, thigh or upper arm) irrespective of the timing of meals. Dose escalation for placebo matched that of liraglutide. Subjects remained on a stable dose of placebo for 56 weeks. Subjects were also on CMS-IBT during the trial.
Period: Overall Study
Arm/Group | Liraglutide 3.0 mg | Placebo
Started | 142 | 140
Completed (Completed without discontinuation of trial product) | 114 | 103
Not Completed | 28 | 37
Not completed — Adverse Event | 12 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 1 | 6
Not completed — Unclassified | 13 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (11.6) | 49 (11.2) | 47.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 116 | 235
  Male | 23 | 24 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 22 | 49
  White | 112 | 115 | 227
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kg] | 108.5 (22.1) | 106.7 (22.0) | 107.6 (22.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Observed mean change in body weight from baseline (week 0) to week 56 was evaluated for two different observation periods. In-trial observation period: the uninterrupted time interval from the date of randomisation until and including the date of the follow-up visit or date of last contact. On-drug observation period: includes all time intervals in which subjects are considered to be on treatment from the date of first trial product administration to 7 days (or 14 days for AEs) after the final trial product administration, excluding potential off-treatment time intervals triggered by at least 7 consecutive missed doses (or 14 consecutive missed doses for AEs).
  The test of superiority of liraglutide to placebo for the treatment policy estimand was tested in a hierarchical manner for the two primary and the consequent 7 confirmatory secondary endpoints presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percent change
  In-trial observation period: number analyzed (Participants) | 141 | 130
  In-trial observation period | -7.4 (7.9) | -4.0 (7.4)
  On-drug observation period: number analyzed (Participants) | 114 | 103
  On-drug observation period | -9.1 (7.4) | -4.8 (7.6)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Treatrment policy estimand. The hypothesis and the alternative are: H: μliraglutide ≥ μplacebo against the alternative HA: μliraglutide < μplacebo. μliraglutide and μplacebo denote the true mean of % weight change for liraglutide 3.0 mg and placebo group, respectively. Week 56 responses were analysed using an analysis of covariance model with treatment, BMI groups, and sex as factors and baseline body weight as covariate; Test type: Superiority — The treatment policy estimand evaluated the treatment effect (liraglutide 3.0 mg vs placebo) at week 56 for all randomised subjects regardless of premature discontinuation of trial product; p = 0.0003, ANCOVA; Missing observations were imputed from the placebo arm based on a jump to reference (x100) multiple imputation approach; Treatment difference = -3.45, 95% CI 2-sided [-5.31 to -1.59] — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Hypothetical estimand. Analysis of on-drug data before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups, and sex as factors and baseline body weight as covariate, all nested within visit; Test type: Other — The hypothetical estimand evaluated the treatment effect (liraglutide 3.0 mg vs placebo) for all randomised subjects assuming that all subjects remained on trial product (on-treatment principle); p = 0.0000, Mixed models repeated measurement (MMRM); Treatment difference = -4.59, 95% CI 2-sided [-6.54 to -2.64] — Liraglutide 3.0 mg - placebo

2. Primary Outcome: Proportion of Subjects Losing at Least 5% of Baseline Body Weight at Week 56
Description: The estimated mean percentage of subjects losing at least 5% of baseline body weight at week 56 is presented. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of participants
  In-trial observation period: number analyzed (Participants) | 141 | 130
  In-trial observation period | 61.47 | 38.82
  On-drug observation period | 64.08 | 38.57
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Treatment policy estimand. Week 56 responses were analysed using a logistic regression model with treatment, BMI groups, and sex as factors and baseline body weight as covariate. Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.53 to 4.14] — Liraglutide 3.0 mg/Placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Hypothetical estimand. Analysis of on-drug before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups, and sex as factors and baseline body weight as covariate, all nested within visit. The MMRM was used to classify responders and analysed with a logistic regression with treatment as the only factor; Test type: Other; p = 0.0000, Mixed models repeated measurement (MMRM); Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.75 to 4.61] — Liraglutide 3.0 mg/placebo

3. Secondary Outcome: Proportion of Subjects Losing More Than 10% of Baseline Body Weight at Week 56
Description: The estimated mean percentage of subjects losing more than 10% of baseline body weight at week 56 is presented. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of participants
  In-trial observation period: number analyzed (Participants) | 141 | 130
  In-trial observation period | 30.45 | 19.75
  On-drug observation period | 33.80 | 19.29
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Treatment policy estimand. Week 56 responses were analysed using a logistic regression model with treatment, BMI groups, and sex as factors and baseline body weight as covariate. Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x10000) imputation approach; Test type: Superiority; p = 0.0469, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.01 to 3.14] — Liraglutide 3.0 mg/Placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.0063, Mixed models repeated measurement (MMRM); Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.24 to 3.69] — Liraglutide 3.0 mg/placebo

4. Secondary Outcome: Proportion of Subjects Losing More Than 15% of Baseline Body Weight at Week 56
Description: The estimated mean percentage of subjects losing more than 15% of baseline body weight at week 56 is presented. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of participants
  In-trial observation period: number analyzed (Participants) | 141 | 130
  In-trial observation period | 18.11 | 8.92
  On-drug observation period | 20.42 | 8.57
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0311, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.08 to 4.74] — Liraglutide 3.0 mg/Placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.0060, Mixed models repeated measurement (MMRM); Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.33 to 5.62] — Liraglutide 3.0 mg/placebo

5. Secondary Outcome: Proportion of Subjects Losing 4% or More of Baseline Body Weight
Description: The estimated mean percentage of subjects losing 4% or more of baseline body weight at week 16 is presented. The endpoint was evaluated for treatment policy estimand (in-trial data).
Time Frame: Week 16
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of participants | 78.73 | 52.70
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Treatment policy estimand. Week 16 responders were analysed using a logistic regression model with treatment, BMI groups, and sex as factors and baseline body weight as covariate. Missing values are considered as non-responders; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.93 to 5.72] — Liraglutide 3.0 mg/placebo

6. Secondary Outcome: Change in Waist Circumference (cm)
Description: Observed mean change from baseline in waist circumference. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
cm
  In-trial observation period: number analyzed (Participants) | 141 | 127
  In-trial observation period | -9.27 (9.22) | -6.91 (8.22)
  On-drug observation period: number analyzed (Participants) | 114 | 103
  On-drug observation period | -10.46 (9.22) | -7.24 (8.67)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach. Week 56 responses were analysed using an analysis of covariance model with treatment, BMI groups, and sex as factors and baseline measurement of endpoint as covariate; Test type: Superiority; p = 0.0063, ANCOVA; treatment difference = -2.72, 95% CI 2-sided [-4.68 to -0.77] — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of on-drug before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups, and sex as factors and baseline measurement of endpoint as covariate, all nested within visit; Test type: Other; p = 0.0020, Mixed model repeated measurements (MMRM); Treatment difference = -3.45, 95% CI 2-sided [-5.62 to -1.28] — Liraglutide 3.0 mg - placebo

7. Secondary Outcome: Change in Short Form-36 (SF-36) v2.0 Acute, Physical Functioning Score
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the subject's overall health-related quality of life (HRQoL).
  SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in SF-36 physical functioning score is presented. A positive change score indicates an improvement since baseline. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Scores on a scale
  In-trial observation period: number analyzed (Participants) | 138 | 121
  In-trial observation period | 3.55 (6.98) | 4.21 (6.85)
  On-drug observation period: number analyzed (Participants) | 114 | 103
  On-drug observation period | 4.03 (6.49) | 4.77 (6.03)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Treatment policy estimand. Analysis of in-trial data with missing observations imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach. Week 56 responses were analysed using an analysis of covariance model with treatment, BMI groups, and sex as factors and baseline measurement of endpoint as covariate; Test type: Superiority; p = 0.8137, ANCOVA; Treatment difference = 0.16, 95% CI 2-sided [-1.19 to 1.52] — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; Hypothetical estimand. Analysis of on-drug before first drug discontinuation date using a mixed model for repeated measurements with treatment, BMI groups, and sex as factors and baseline measurement of endpoint as covariate, all nested within visit; Test type: Other; p = 0.8053, Mixed model repeated measurements (MMRM); Treatment difference = 0.16, 95% CI 2-sided [-1.12 to 1.43] — Liraglutide 3.0 mg- placebo

8. Secondary Outcome: Change in IWQoL-Lite for CT, Physical Function Domain (5-items) Score
Description: Observed mean change in Impact of Weight on Quality of Life-Lite for Clinical Trials Version (IWQoL-Lite for CT ) score. IWQoL-Lite for CT (Weight on Quality of Life-Lite for Clinical Trial Version) is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life.
  The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Scores on a scale
  In-trial observation period: number analyzed (Participants) | 138 | 121
  In-trial observation period | 13.5 (21.4) | 15.5 (23.0)
  On-drug observation period: number analyzed (Participants) | 114 | 103
  On-drug observation period | 15.2 (21.4) | 17.5 (21.4)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Superiority was not tested as part of confirmatory testing strategy; p = 0.6916, ANCOVA; Treatment difference = 0.87, 95% CI 2-sided [-3.41 to 5.14] — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.5572, Mixed models repeated measurements (MMRM; treatment difference = 1.25, 95% CI 2-sided [-2.95 to 5.45] — Liraglutide 3.0 mg - placebo

9. Secondary Outcome: Change in Six Minutes Walking Distance Test (6MWT)
Description: Observed mean change from baseline in 6 minutes walking distance test. The 6MWT is a common test of functional exercise capacity that assesses the distance a subject can walk in 6 minutes. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
meter
  In-trial observation period: number analyzed (Participants) | 135 | 116
  In-trial observation period | 47 (59) | 49 (69)
  On-drug observation period: number analyzed (Participants) | 112 | 101
  On-drug observation period | 53 (61) | 51 (69)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Superiority was not tested as part of confirmatory testing strategy; p = 0.6986, ANCOVA; Treatment difference = 3.12, 95% CI 2-sided [-12.68 to 18.92] — Liraglutide 3.0 mg - placebo
Statistical Analysis 2: Comparison: Liraglutide 3.0 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.3700, Mixed model repeated measurements (MMRM); Treatment difference = 7.66, 95% CI 2-sided [-9.15 to 24.48] — Liraglutide 3.0 mg - placebo

10. Secondary Outcome: Change From Baseline in HbA1c (%)
Description: Observed mean change from baseline to week 56 in glycosylated haemoglobin (HbA1c). Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage | -0.2 (0.3) | -0.1 (0.2)

11. Secondary Outcome: Change From Baseline in FPG (mg/dL)
Description: Observed mean change from baseline (week 0) in fasting plasma glucose (FPG). Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mg/dL | -4.04 (9.59) | -0.28 (11.46)

12. Secondary Outcome: Change From Baseline sBP (mmHg)
Description: Observed mean change in systolic blood pressure from baseline to week 56.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmHg | -2 (14) | -1 (13)

13. Secondary Outcome: Change From Baseline dBP (mmHg)
Description: Observed mean change from baseline (week 0) to week 56 in diastolic blood pressure (dBP). Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmHg | -1 (11) | -1 (10)

14. Secondary Outcome: Change From Baseline in Lipids -Total Cholesterol
Description: Observed mean change from baseline (week 0) to week 56 in total cholesterol (TC). Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.01 (0.59) | 0.00 (0.77)

15. Secondary Outcome: Change From Baseline in Lipids - LDL Cholesterol
Description: Observed mean change from baseline in low density cholesterol (LDL) from baseline (week 0) to week 56. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.01 (0.52) | -0.01 (0.64)

16. Secondary Outcome: Change From Baseline in Lipids - HDL Cholesterol
Description: Observed mean change from baseline in high density (HDL) cholesterol from baseline (week 0) to week 56. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | 0.06 (0.19) | 0.02 (0.22)

17. Secondary Outcome: Change From Baseline in Lipids - VLDL Cholesterol
Description: Observed mean change from baseline in very low density cholesterol (VLDL) from baseline (week 0) to week 56. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.06 (0.31) | -0.01 (0.26)

18. Secondary Outcome: Change From Baseline in Lipids - TG
Description: Observed mean change from baseline in triglyceride (TG) from baseline (week 0) to week 56. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.19 (1.04) | -0.01 (0.58)

19. Secondary Outcome: Change From Baseline in Lipids - FFA
Description: Observed mean change from baseline in free fatty acids (FFA) from baseline (week 0) to week 56. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.07 (0.28) | -0.06 (0.31)

20. Secondary Outcome: Change in Short Form-36 v2.0 Acute (SF-36) (Subdomains)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the subject's overall health-related quality of life (HRQoL).
  SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in in the sub-domain scores is presented. A positive change score indicates an improvement since baseline. Results are evaluated based on in-trial data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
scores on a scale
  Bodily Pain: number analyzed (Participants) | 138 | 121
  Bodily Pain | 0.67 (7.61) | 1.21 (8.88)
  General Health Perception: number analyzed (Participants) | 138 | 121
  General Health Perception | 1.89 (6.31) | 1.08 (6.62)
  Mental Health: number analyzed (Participants) | 138 | 121
  Mental Health | -0.93 (7.80) | -0.68 (6.89)
  Role Lim Emotion Prob: number analyzed (Participants) | 138 | 121
  Role Lim Emotion Prob | -1.27 (7.72) | -2.21 (8.59)
  Role Lim. Phy Health: number analyzed (Participants) | 138 | 121
  Role Lim. Phy Health | 2.01 (6.55) | 2.11 (7.68)
  Social Functioning: number analyzed (Participants) | 138 | 121
  Social Functioning | 1.22 (8.69) | -0.45 (9.61)
  Vitality: number analyzed (Participants) | 138 | 121
  Vitality | 2.64 (8.99) | 2.43 (7.78)

21. Secondary Outcome: Change in Short Form-36 v2.0 Acute (SF-36) (Physical Component Summary (PCS))
Description: Observed mean change from baseline (week 0) to week 56 in short form 36 v2.0 acute domain physical component summary (PCS). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in SF-36 physical component summary (PCS) score is presented. A positive change score indicates an improvement since baseline. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
scores on a scale | 3.41 (6.65) | 3.83 (7.22)

22. Secondary Outcome: Change in Short Form-36 v2.0 Acute (SF-36) (Mental Component Summary (MCS)
Description: Observed mean change from baseline (week 0) to week 56 in short form 36 v2.0 acute domain mental component summary (MCS). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in SF-36 mental component summary is presented. A positive change score indicates an improvement since baseline. The endpoint was evaluated based on in-trial data and on-drug data.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
scores on a scale | -1.22 (8.74) | -2.20 (8.11)

23. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT): Pain/Discomfort Domain Score
Description: Observed mean change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT) domain pain and discomfort. IWQoL-Lite for CT (Weight on Quality of Life-Lite for Clinical Trial Version) is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
scores on a scale | 10.1 (21.2) | 8.6 (23.1)

24. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT): Psychosocial Domain Score
Description: Observed mean change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT) psychosocial domain. IWQoL-Lite for CT (Weight on Quality of Life-Lite for Clinical Trial Version) is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
score | 13.5 (20.3) | 12.4 (21.8)

25. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite for Clinical Trial Version (IWQoL-Lite for CT): Total Score
Description: Observed mean change from baseline (week 0) to week 56 in IWQoL-Lite for CT total score. IWQoL-Lite for CT (Weight on Quality of Life-Lite for Clinical Trial Version) is a modified version of an instrument designed to assess weight-related quality of life. The scores ranged between 0-100 where higher scores indicated a better quality of life. A positive change score indicates an improvement since baseline. Results based on FAS in-trial data is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
scores on a scale | 13.2 (18.5) | 12.8 (20.7)

26. Secondary Outcome: Change in Weight Related Sign and Symptom (WRSS) Measure, Total Score
Description: Observed mean change from baseline (week 0) to week 56 in WRSS measure, total score. The WRSS measures the presence and bothersome associated with weight-related symptoms.
  The WRSS questionnaire was not validated until after database lock. Therefore the total score couldn't be calculated and the supportive secondary endpoint "Weight related sign and symptom (WRSS) measure, total score" couldn't be analysed.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Score on a scale | NA (NA) — The WRSS questionnaire was not validated until after database lock. Therefore the total score couldn't be calculated and the supportive secondary endpoint "Weight related sign and symptom (WRSS) measure, total score" couldn't be analysed. | NA (NA) — The WRSS questionnaire was not validated until after database lock. Therefore the total score couldn't be calculated and the supportive secondary endpoint "Weight related sign and symptom (WRSS) measure, total score" couldn't be analysed.

27. Secondary Outcome: Subjects Who After 56 Weeks Achieve (Yes/no): ≥ 4.3 T-score Points Increase From Baseline in SF-36 Physical Functioning Score
Description: Percentage of subjects who achieved ≥ 4.3 T-score points increase from baseline in SF-36 physical functioning score at week 56 is presented. Results based on FAS in-trial data is presented.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of participants | 38.7 | 37.9

28. Secondary Outcome: Subjects Who After 56 Weeks Achieve (Yes/no): ≥ 3.8 T-score Points Increase From Baseline in SF-36 Physical Component Score
Description: Percentage of subjects who achieved ≥ 3.8 T-score points increase from baseline in SF-36 physical component score at week 56 is presented. Results based on FAS in-trial data is presented.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Percentage of participants | 43.7 | 41.4

29. Secondary Outcome: Subjects Who After 56 Weeks Achieve (Yes/no): ≥ 4.6 T-score Points Increase From Baseline in SF-36 Mental Component Score
Description: Percentage of subjects who achieved ≥ 4.6 T-score points increase from baseline in SF-36 mental component score at week 56 is presented. Results based on FAS in-trial data is presented.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Percentage of participants | 20.4 | 9.3

30. Secondary Outcome: Responder Definition Value for IWQoL-Lite for CT Physical Function Domain (5-items) Score
Description: Responder definition value for IWQoL-Lite for CT physical function domain (5-items) score' was defined as '≥ 20 responder definition value for IWQoL-Lite for CT physical function domain (5-items) score. Percentage of subjects considered IWQoL-Lite for CT physical function domain score responders (increase of ≥20 points) at week 56 is presented. Results based on FAS in-trial data is presented.
Time Frame: Week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
Percentage of participants | 37.3 | 34.3

31. Secondary Outcome: Number of Weeks (Completed Calendar Weeks) From Randomisation to Week 56 Adherent to Trial Product
Description: Adherence to trial product is assessed regularly at CMS-IBT visits. The number of weeks from randomisation to week 56, adherent to trial product is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
weeks | 49.5 (14.0) | 46.8 (16.1)

32. Secondary Outcome: Number of Weeks (Completed Calendar Weeks) From Randomisation to Week 56 Adherent to Caloric Diet
Description: Adherence to caloric diet is assessed regularly at CMS-IBT visits. The number of weeks from randomisation to week 56, adherent to caloric diet is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
weeks | 38.4 (16.0) | 36.1 (17.3)

33. Secondary Outcome: Number of Weeks (Completed Calendar Weeks) From Randomisation to Week 56 Adherent to Physical Activity
Description: Adherence to physical activity is assessed regularly at CMS-IBT visits. The number of weeks from randomisation to week 56, adherent to physical activity is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
weeks | 29.0 (17.1) | 30.0 (17.2)

34. Secondary Outcome: Number of Weeks (Completed Calendar Weeks) From Randomisation to Week 56 Adherent to Caloric Diet and Physical Activity
Description: Adherence to caloric diet and physical activity is assessed regularly at CMS-IBT visits. The number of weeks from randomisation to week 56, adherent to caloric diet and physical activity is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
weeks | 24.0 (16.0) | 24.5 (15.7)

35. Secondary Outcome: Number of Weeks (Completed Calendar Weeks) From Randomisation to Week 56 Adherent to Caloric Diet, Physical Activity and Trial Product
Description: Adherence to caloric diet, physical activity and trial product is assessed regularly at CMS-IBT visits. The number of weeks from randomisation to week 56, adherent to caloric diet, physical activity and trial product is presented.
Time Frame: Week 0, week 56
Population: Full analysis set included all randomised subjects. "Number analysed"=subjects with available data.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
weeks | 22.9 (16.1) | 24.0 (15.9)

36. Secondary Outcome: AEs From Randomisation Until and Including the Follow-up Period
Description: Number of adverse events from randomisation to until the end of the post-treatment follow-up period (30 days). Results based on SAS on-drug data is presented.
Time Frame: Week 0 to week 56+30 days
Population: Safety analysis set included all randomised subjects exposed to at least one dose of trial drug. "Number analysed"=subjects with available data.
Measure: Number; unit: events
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
events | 867 | 601

37. Secondary Outcome: Change in Physical Examination
Description: Observed change from baseline to week 56 in physical examination are categorised under parameters namely abdomen, gastrointestinal system, cardiovascular system, central and peripheral nervous system, general appearence, head, ears, eyes, nose, throat and neck, lymph node palpation, musculoskeletal system, respiratory system, skin and thyroid gland. The percentage of subjects assessed as normal, abnormal not clinically significant and abnormal clinically significant at baseline and week 56 is presented.
Time Frame: Week 1, week 56
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
participants
  Abdomen (week -1) Normal | 108 | 121
  Abdomen (week -1) Abnormal, NCS | 34 | 19
  Abdomen (week -1) Abnormal CS | 0 | 0
  Abdomen (week 56) Normal: number analyzed (Participants) | 139 | 122
  Abdomen (week 56) Normal | 114 | 108
  Abdomen (week 56) Abnormal, NCS: number analyzed (Participants) | 139 | 122
  Abdomen (week 56) Abnormal, NCS | 25 | 12
  Abdomen (week 56) Abnormal, CS: number analyzed (Participants) | 139 | 122
  Abdomen (week 56) Abnormal, CS | 0 | 2
  Gastrointestinal System (week -1) Normal | 130 | 129
  Gastrointestinal System (week -1) Abnormal NCS | 12 | 11
  Gastrointestinal System (week -1) Abnormal CS | 0 | 0
  Gastrointestinal System (week 56) Normal: number analyzed (Participants) | 139 | 122
  Gastrointestinal System (week 56) Normal | 132 | 116
  Gastrointestinal System (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Gastrointestinal System (week 56) Abnormal NCS | 7 | 6
  Gastrointestinal System (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Gastrointestinal System (week 56) Abnormal CS | 0 | 0
  Cardiovascular System (week-1) Normal | 136 | 127
  Cardiovascular System (week-1) Abnormal NCS | 6 | 13
  Cardiovascular System (week-1) Abnormal CS | 0 | 0
  Cardiovascular System (week 56) Normal: number analyzed (Participants) | 139 | 122
  Cardiovascular System (week 56) Normal | 138 | 116
  Cardiovascular System (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Cardiovascular System (week 56) Abnormal NCS | 1 | 5
  Cardiovascular System (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Cardiovascular System (week 56) Abnormal CS | 0 | 1
  Nervous System (week -1) Normal | 135 | 127
  Nervous System (week -1) Abnormal NCS | 5 | 6
  Nervous System (week -1) Abnormal CS | 2 | 7
  Nervous System (week 56) Normal: number analyzed (Participants) | 139 | 122
  Nervous System (week 56) Normal | 132 | 112
  Nervous System (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Nervous System (week 56) Abnormal NCS | 6 | 9
  Nervous System (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Nervous System (week 56) Abnormal CS | 1 | 1
  General Appearance (week -1) Normal | 118 | 123
  General Appearance (week -1) Abnormal NCS | 24 | 17
  General Appearance (week -1) Abnormal CS | 0 | 0
  General Appearance (week 56) Normal: number analyzed (Participants) | 139 | 122
  General Appearance (week 56) Normal | 122 | 112
  General Appearance (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  General Appearance (week 56) Abnormal NCS | 17 | 10
  General Appearance (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  General Appearance (week 56) Abnormal CS | 0 | 0
  Head, ENTand Neck (week -1) Normal | 129 | 128
  Head, ENTand Neck (week -1) Abnormal NCS | 13 | 12
  Head, ENTand Neck (week -1) Abnormal CS | 0 | 0
  Head, ENTand Neck (week 56) Normal: number analyzed (Participants) | 139 | 122
  Head, ENTand Neck (week 56) Normal | 126 | 115
  Head, ENTand Neck (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Head, ENTand Neck (week 56) Abnormal NCS | 13 | 7
  Head, ENTand Neck (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Head, ENTand Neck (week 56) Abnormal CS | 0 | 0
  Lymph Node Palpation (week -1) Normal | 142 | 140
  Lymph Node Palpation (week -1) Abnormal NCS | 0 | 0
  Lymph Node Palpation (week -1) Abnormal CS | 0 | 0
  Lymph Node Palpation (week 56) Normal: number analyzed (Participants) | 139 | 122
  Lymph Node Palpation (week 56) Normal | 139 | 121
  Lymph Node Palpation (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Lymph Node Palpation (week 56) Abnormal NCS | 0 | 0
  Lymph Node Palpation (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Lymph Node Palpation (week 56) Abnormal CS | 0 | 1
  Musculoskeletal System (week -1) Normal | 131 | 128
  Musculoskeletal System (week -1) Abnormal NCS | 11 | 12
  Musculoskeletal System (week -1) Abnormal CS | 0 | 0
  Musculoskeletal System (week 56) Normal: number analyzed (Participants) | 139 | 122
  Musculoskeletal System (week 56) Normal | 130 | 112
  Musculoskeletal System (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Musculoskeletal System (week 56) Abnormal NCS | 9 | 9
  Musculoskeletal System (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Musculoskeletal System (week 56) Abnormal CS | 0 | 1
  Respiratory System (week -1) Normal | 140 | 138
  Respiratory System (week -1) Abnormal NCS | 2 | 2
  Respiratory System (week -1) Abnormal CS | 0 | 0
  Respiratory System (week 56) Normal: number analyzed (Participants) | 139 | 122
  Respiratory System (week 56) Normal | 138 | 120
  Respiratory System (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Respiratory System (week 56) Abnormal NCS | 1 | 2
  Respiratory System (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Respiratory System (week 56) Abnormal CS | 0 | 0
  Skin (week -1) Normal | 116 | 114
  Skin (week -1) Abnormal NCS | 26 | 24
  Skin (week -1) Abnormal CS | 1 | 0
  Skin (week 56) Normal: number analyzed (Participants) | 139 | 122
  Skin (week 56) Normal | 117 | 98
  Skin (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Skin (week 56) Abnormal NCS | 21 | 24
  Skin (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Skin (week 56) Abnormal CS | 1 | 0
  Thyroid Gland (week -1) Normal | 138 | 138
  Thyroid Gland (week -1) Abnormal NCS | 4 | 2
  Thyroid Gland (week -1) Abnormal CS | 0 | 0
  Thyroid Gland (week 56) Normal: number analyzed (Participants) | 139 | 122
  Thyroid Gland (week 56) Normal | 136 | 120
  Thyroid Gland (week 56) Abnormal NCS: number analyzed (Participants) | 139 | 122
  Thyroid Gland (week 56) Abnormal NCS | 3 | 2
  Thyroid Gland (week 56) Abnormal CS: number analyzed (Participants) | 139 | 122
  Thyroid Gland (week 56) Abnormal CS | 0 | 0

38. Secondary Outcome: Change in Resting Pulse
Description: Observed mean change in pulse rate measured at resting position is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
beats/min | 2 (10) | 1 (10)

39. Secondary Outcome: Change in ECG
Description: The ECGs were interpreted by the investigator at baseline (week -1) and week 56 and categorised as normal, abnormal NCS or abnormal CS. Number of subjects in each ECG category at baseline and week 56 are presented.
Time Frame: Week -1, week 56
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
participants
  Normal (week -1) | 100 | 91
  Abnormal NCS (week -1) | 41 | 49
  Abnormal CS (week -1) | 1 | 0
  Normal (week 56): number analyzed (Participants) | 138 | 124
  Normal (week 56) | 102 | 81
  Abnormal NCS (week 56): number analyzed (Participants) | 138 | 124
  Abnormal NCS (week 56) | 36 | 42
  Abnormal CS (week 56): number analyzed (Participants) | 138 | 124
  Abnormal CS (week 56) | 0 | 1

40. Secondary Outcome: Change in Laboratory Measurements: Haematology (Haemoglobin Blood)
Description: Observed mean change from baseline in haematological parameter blood haemoglobin.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L | -0.2 (0.5) | -0.1 (0.6)

41. Secondary Outcome: Change in Laboratory Measurements: Haematology (Haematocrit Blood)
Description: Observed mean change from baseline in haematological parameter blood haematocrit. Haematocrit is presented as the percentage of red blood cells in total blood. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
percentage of red blood cells | -1.5 (2.3) | -0.9 (2.6)

42. Secondary Outcome: Change in Laboratory Measurements: Haematology (Erythrocytes)
Description: Observed mean change from baseline in haematological parameter - erythrocytes.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
10^12 cells/L | -0.11 (0.25) | -0.08 (0.25)

43. Secondary Outcome: Change in Laboratory Measurements: Haematology (Thrombocytes and Leukocytes)
Description: Observed mean change from baseline in haematological parameters - thrombocytss and leukocytes.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
10^9 cells/L
  Thrombocytes: number analyzed (Participants) | 109 | 101
  Thrombocytes | 4 (30) | 0 (36)
  Leukocytes: number analyzed (Participants) | 110 | 101
  Leukocytes | -0.14 (1.53) | -0.11 (1.20)

44. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Albumin)
Description: Observed mean change from baseline in biochemical parameter - albumin. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
g/L | -0.1 (0.2) | -0.1 (0.2)

45. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Alkaline Phosphatase, Alanine Aminotransferase, Amylase, Aspartate Aminotransferase and Lipase)
Description: Observed mean change from baseline in biochemical parameters - alkaline phosphatase, alanine aminotransferase, amylase, aspartate aminotransferase and lipase. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
U/L
  Alkaline Phosphatase: number analyzed (Participants) | 111 | 103
  Alkaline Phosphatase | -2 (12) | -1 (13)
  Alanine Aminotransferase: number analyzed (Participants) | 111 | 103
  Alanine Aminotransferase | -5 (14) | -4 (16)
  Amylase: number analyzed (Participants) | 111 | 103
  Amylase | 4 (10) | 1 (13)
  Aspartate aminotransferase: number analyzed (Participants) | 110 | 103
  Aspartate aminotransferase | -3 (10) | -2 (12)
  Lipase: number analyzed (Participants) | 111 | 103
  Lipase | 7 (18) | 2 (22)

46. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Bilirubin and Creatinine)
Description: Observed mean change from baseline in biochemical parameters - bilirubin and creatinine. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
umol/L
  Bilirubin: number analyzed (Participants) | 111 | 103
  Bilirubin | 1.1 (3.2) | 1.0 (3.2)
  Creatinine: number analyzed (Participants) | 111 | 103
  Creatinine | -1.8 (7.9) | -1.4 (6.1)

47. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Total Calcium, Pottassium, Sodium and Urea)
Description: Observed mean change from baseline in biochemical parameters - total calcium, pottassium, sodium and urea. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mmol/L
  Total Calcium: number analyzed (Participants) | 111 | 103
  Total Calcium | 0.01 (0.10) | 0.01 (0.09)
  Potassium: number analyzed (Participants) | 111 | 103
  Potassium | -0.0 (0.5) | -0.0 (0.4)
  Sodium: number analyzed (Participants) | 111 | 103
  Sodium | -0.0 (2) | -0 (2)
  Urea: number analyzed (Participants) | 111 | 103
  Urea | 0.0 (1.2) | 0.2 (1.2)

48. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (C-reactive Protein and Uric Acid)
Description: Observed mean change from baseline in biochemical parameters - high sensitive c-reactive protein and uric acid. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mg/dL
  High sensitive c-reactive protein: number analyzed (Participants) | 111 | 103
  High sensitive c-reactive protein | -2.51 (4.67) | -0.85 (8.96)
  Uric acid: number analyzed (Participants) | 111 | 103
  Uric acid | -0.6 (0.9) | -0.3 (0.9)

49. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Glomerular Filtration Rate, Serum)
Description: Observed mean change from baseline in biochemical parameters - estimated glomerular filtration rate. Serum GFR is estimated using MDRD formula . Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mL/min/1.73m^2 | 2 (11) | 2 (9)

50. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Calcitonin)
Description: Observed mean change from baseline in biochemical parameter - calcitonin. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
ng/L | 0.2 (0.8) | 0.1 (0.8)

51. Secondary Outcome: Change in Laboratory Measurements: Biochemistry (Thyroid Stimulating Hormone)
Description: Observed mean change from baseline in biochemical parameters - thyroid stimulating hormone. Results based on SAS on-drug data is presented.
Time Frame: Week 0, week 56
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 142 | 140
mIU/L | -0.2313 (1.0366) | 0.2685 (3.6814)

ADVERSE EVENTS:
Time Frame: From the date of first dose of trial product (week 0) to end of treatment (week 56) + post treatment follow-up of 30 days.
Description: Evaluation of safety was based on safety analysis set (SAS) which comprised of all randomised subjects who received at least one dose of trial product.
  AEs with onset during the on-drug observation period (the period when subjects were exposed to trial product) were considered treatment-emergent.
Groups:
- Lira 3.0 mg: Subjects received liraglutide 3.0 mg once daily by subcutaneous injection (in the abdomen, thigh or upper arm) irrespective of the timing of meals. Subjects received 0.6 mg liraglutide during the first week. The dose was escalated in weekly increments of 0.6 mg until they reached a maintenance dose of 3.0 mg after 4 weeks. The treatment period was 56 weeks. Subjects were also on CMS-IBT during the trial.
Arm/Group | Lira 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/140
Serious Adverse Events (participants affected / at risk) | 6/142 | 2/140
Other Adverse Events (participants affected / at risk) | 124/142 | 101/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 3.0 mg (N=142) | Placebo (N=140)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 3.0 mg (N=142) | Placebo (N=140)
Abdominal discomfort (Gastrointestinal disorders) | 8 (9) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 16 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 13 (14)
Constipation (Gastrointestinal disorders) | 43 (57) | 26 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 31 (47) | 23 (26)
Dizziness (Nervous system disorders) | 9 (10) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 8 (13) | 3 (3)
Fatigue (General disorders) | 13 (15) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 3 (5) | 9 (9)
Headache (Nervous system disorders) | 20 (23) | 13 (29)
Influenza (Infections and infestations) | 5 (5) | 13 (13)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6) | 9 (9)
Migraine (Nervous system disorders) | 3 (3) | 9 (12)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 7 (8)
Nasopharyngitis (Infections and infestations) | 13 (17) | 9 (13)
Nausea (Gastrointestinal disorders) | 68 (102) | 25 (33)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8)
Sinusitis (Infections and infestations) | 9 (10) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 32 (38) | 15 (17)
Urinary tract infection (Infections and infestations) | 8 (15) | 3 (3)
Vomiting (Gastrointestinal disorders) | 33 (47) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02963935/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02963935/SAP_001.pdf